CLINICAL TRIAL: NCT03610282
Title: Electroencephalogram Study of Intravenous Methylphenidate-Induced Emergence From Propofol Sedation
Brief Title: EEG Study of IV Methylphenidate-Induced Emergence From Propofol Sedation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We have decided to withdraw the study prior to enrollment of the first participant in order to pursue other research studies.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ken Solt, MD, Associate Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018P001421
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia
Keywords: Propofol; Methylphenidate; Ritalin; Anesthetics; Anesthetics, Intravenous; Molecular Mechanisms of Pharmacological Action; Anesthetics, General; Neurotransmitter Agents; Physiological Effects of Drugs
MeSH Terms: interventions — Methylphenidate; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EEG Dynamics (Experimental): EEG data will be collected on patients receiving propofol and IV methylphenidate together.
  Interventions: Drug: IV Methylphenidate; Drug: Propofol
- Propofol EEG Dynamics (Placebo Comparator): EEG data will be collected on patients receiving propofol and a saline placebo.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: IV Methylphenidate — Subjects will receive a bolus of IV methylphenidate during propofol infusion at one of the study visits.
  Other Names: Ritalin
  Arms: EEG Dynamics
Drug: Propofol — Subjects will received propofol for up to 100 minutes.

SUMMARY:
The investigators are performing this research study to find out if intravenous (IV) methylphenidate (commonly known as Ritalin) can help people recover faster from propofol sedation. The investigators also want to know how IV methylphenidate acts in the brain and whether IV methylphenidate is safe to take with an anesthetic (a drug or agent used to decrease or eliminate the feeling of pain by causing unconsciousness) without causing too many side effects. The brain's electrical activity will be studied and recorded using a machine called an electroencephalogram (EEG).

DETAILED DESCRIPTION:
During this research study, participants will receive propofol, and propofol and IV methylphenidate together, at a high enough dose to achieve unconsciousness (make study participants "fall asleep"). During one visit participants will receive propofol and a saline placebo; during another visit participants will be given both propofol and IV methylphenidate together. The investigators will record EEG the entire time, The investigators will also ask some questions related to cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 45
* Normal body weight and habitus, BMI ≤ 30
* Non-smoker
* No history of taking stimulants
* American Society of Anesthesiologists (ASA) physical status classification P1

Exclusion Criteria:

• Chronic health conditions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in multitaper spectral estimates of EEG power during a continuous infusion of propofol. | Up to 100 minutes
  Change from baseline in multitaper spectral estimates of EEG power associated with the administration of IV methylphenidate.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Solt, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States